CLINICAL TRIAL: NCT06148493
Title: Real-World Usage of Asciminib Among Patients With Chronic Myeloid Leukemia in Chronic Phase in the United States Using a Large Claims Database
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CABL001A0US01
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Chronic Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This was a retrospective descriptive analysis of health care claims data using the IQVIA open source medical and pharmacy claims databases. Patients were grouped into one of two cohorts depending on the index medication.

All patients with at least 1 pharmacy claim for asciminib occurring between 01 January 2021 and 30 April 2022 in (Phase 1) were grouped into the asciminib cohort. A data refresh was conducted (Phase 1 refresh) and all patients with at least 1 pharmacy claim for asciminib occurring between 01 January 2021 and 29 August 2022 were included in the asciminib cohort. Patients were required to have at least 6 months of continuous data availability prior to the start of treatment and were followed from the start of treatment until the end of available follow-up. The end of available follow up in open source data was defined as 1) last claim date in medical or pharmacy data, OR 2) last day of index pharmacy stability, OR 3) end of study period, whichever came first. While no post-index data availability were required in Phase 1, a subgroup analysis was conducted in patients with at least 3 and 6 months of available follow-up after the index date in Phase 1 refresh.

In Phase 2 of the study, patients with no exposure to asciminib and with at least 1 pharmacy claim for imatinib mesylate, dasatinib, nilotinib, bosutinib or ponatinib were indexed to the first new tyrosine kinase inhibitor (TKI) observed between 01 January 2021 and 29 August 2022 and grouped into the other TKI cohort. The index date was the initiation date of the index medication. Patients were required to have linkage to the open-source medical claims database and at least 3 months of available follow-up after the index date.

ELIGIBILITY:
Inclusion criteria:

Patients meeting the below inclusion criteria were included in the study.

* Patients with ≥ 1 claim for asciminib (asciminib cohort) or another third-line TKI used to treat CML (imatinib mesylate, dasatinib, nilotinib, bosutinib, ponatinib) in the open-source pharmacy claims database occurring during the index period. All patients with at least one claim for asciminib during the index window were placed into the asciminib cohort and the index date was date of the first asciminib claim. Patients with no claims for asciminib were placed in the other TKI cohort. These patients were indexed on their third-line TKI (i.e., 2 prior TKIs must have been observed at any time prior to the index date) and the index date was the date of the first claim observed during the index period.
* Age ≥ 18 years on the index date.
* Patients with ≥ 6 months of continuous pre-index data availability. This was defined as:

  * The index pharmacy was a stable provider for each of the 6 months prior to the index date; and
  * The patient had at least 1 claim (for any drug) in the open-source pharmacy claims database more than 6 months prior to the index date.

In Phase 2, patients were required to meet the following criteria:

* Patients with linkage to the open-source medical claims database.
* Patients with ≥ 3 months of post-index data availability. Post-index data availability was defined as:

  * The index pharmacy was a stable provider for each of the 3 months after the index date; and
  * The patient had at least 1 claim (for any drug) in the open-source pharmacy claims database more than 3 months after the index date.

Exclusion criteria:

• Patients with data quality issues, defined as missing or invalid age. In order to retain the maximum sample of asciminib patients for the primary objectives, no additional exclusion criteria were applied.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study
Sampling Method: Non-Probability Sample
Enrollment: 425 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Age of patients | Baseline
Sex of patients | Baseline
Geographic region of patients | Baseline
Payer type for prescriptions | Baseline
Total duration of available follow-up | Up to 6 months
Number of patients with chronic myeloid leukemia (CML) diagnosis | Up to 6 months
Specialty of prescribing physician | Up to 6 months
Number of patients with T315I mutation proxy | Up to 6 months
National Cancer Institute (NCI) comorbidity index for patients | Up to 6 months
  The NCI comorbidity index score range is 0, 1 to 2, 2 to 3, and 3+, with higher scores indicating more comorbidity.
Number of patients with comorbidities | Up to 6 months
Pre-index medication use | Up to 6 months
Number of patients with any prior TKI use | Up to 6 months
Number of patients with any prior non-TKI CML treatment | Up to 6 months
Starting dose of index medication | Up to 6 months
Total day supply of index medication | Up to 6 months
Number of prescriptions of index medication | Up to 6 months
Number of patients still on index therapy at the end of Month 3 post-index | Up to 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States